CLINICAL TRIAL: NCT03789890
Title: An Open-label, Single Group Study to Evaluate the Effect of Repeated Oral Administration of Itraconazole (ITZ) on the Single Oral Dose Pharmacokinetics of BAY1902607 in Healthy Male Participants
Brief Title: Study to Learn More About the Effect of Itraconazole (ITZ) Given Repeatedly by Mouth on the Way How the Study Drug BAY1902607 Given One Time by Mouth Acts in the Human Body of Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19431; 2018-003212-50 (EudraCT Number)
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Drug Interactions
Keywords: Drug-drug interaction; Itraconazole (ITZ); Cytochrom P450 3A4 (CYP3A4) metabolism; P2X3-inhibitor
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy men (Experimental): Healthy male adults from Germany receiving BAY1902607 during study period 1 (length = 6 days) and BAY1902607 + Itraconazole during study period 2 (length = 15 days), separated by a washout phase.
  Interventions: Drug: BAY1902607; Drug: Itraconazole

INTERVENTIONS:
Drug: BAY1902607 — BAY1902607 is administered once orally as tablets on Day 2 of study period 1 and on Day 4 of study period 2.
Drug: Itraconazole — Itraconazole is administered at a dose of 200 mg once a day (oral solution of 10 mg mL-1) on Day 1 to Day 14 of study period 2.

SUMMARY:
BAY1902607 is a new type of drug under clinical development for different conditions including the treatment of endometriosis, i.e. a condition where the tissue that usually grows inside the womb grows outside of the womb.

Itraconazole (ITZ) is an approved drug often used for the treatment of fungal infections and possibly inhibits the breakdown of BAY1902607. In this clinical study, BAY1902607 is given alone by mouth or in combination with ITZ. Researchers want to learn more how quickly and to what extent the study drug BAY1902607 given by mouth to healthy male participants is absorbed by the human body, reaches the blood stream and is excreted again. In addition they want to find out whether the elimination of the study drug BAY1902607 is influenced by ITZ given at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male adults
* Body mass index ≥ 18 and ≤ 30.0 kg/m²
* Body weight ≥ 50 kg

Exclusion Criteria:

* Known or suspected allergy or hypersensitivity to BAY1902607, itraconazole or any of their excipients
* Contraindications to itraconazole (symptoms or history of ventricular dysfunction, heart failure, liver disease).
* Any use of systemic or topically active medication or herbal remedies, prescription or non-prescription, within 1 week prior to the first drug administration or during the trial until follow-up (occasional use of ibuprofen is permissible). Particularly, this includes drugs that might affect the pharmacokinetics (PK) of BAY1902607, e.g. laxatives, loperamide, metoclopramide, antacids, H2-receptor antagonists, CYP3A4 inhibitors or inducers.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Cmax of BAY1902607 | -0.5 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36, 48, 96 hours after drug
  Maximum concentration of BAY1902607 in blood
Cmax of BAY1902607 with itraconazole | -1.5 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours after BAY1902607
  Maximum concentration of BAY1902607 in blood with concomitant administration of itraconazole
AUC of BAY1902607 | -0.5 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36, 48, 96 hours after drug
  Area under the concentration versus time curve of BAY1902607 (time from 0 to 96 hours) after single dose
AUC of BAY1902607 with itraconazole | -1.5 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours after BAY1902607
  Area under the concentration versus time curve (time from 0 to 264 hours) after single dose of BAY1902607 and concomitant administration of itraconazole

OTHER OUTCOMES:
Number of participants with treatment-emergent adverse events | Up to 5 weeks
Intensity of treatment-emergent adverse events | Up to 5 weeks
  Adverse events will be assigned to one of three categories: mild (easily tolerated and no interference with everyday activities), moderate (sufficient discomfort and interferes with everyday activities) & severe (prevents normal everyday activities).

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.